CLINICAL TRIAL: NCT03360513
Title: Determining Shapes and Dimensions of Dental Arches for the Use in Lingual Technique.
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Mario Cappellette Jr , PhD,DDS, Orientor, Federal University of São Paulo
Other Study IDs: FUSãoPaulo15
Record Dates: First submitted 2017-11-28; First posted 2017-12-04 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Dental Arch Relationship Anomaly
Keywords: Orthodontics; Dental arch; Orthodontic appliance design.

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — the study sample comprised 70 caucasian brazilian individuals with normal occlusion and at least four of Andrew's six keys.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- general group: Comprised 70 caucasian Brazilian individuals with normal occlusion and at least four of Andrew's six keys.
  Interventions: Other: general group

INTERVENTIONS:
Other: general group — The sample comprised maxillary and mandibular dental casts of 70 Caucasian Brazilian individuals (28 men and 42 women) with an average age of 16.4 years, all of which had natural normal occlusion with at least four of the six keys to normal occlusion. 14 The first item of the first key was considered essential for sample selection(Angle Class I molar relationship). Another inclusion criterion was that individuals should be at least 15 years of age with no odontogenic abnormalities and all permanent teeth in occlusion.

SUMMARY:
This study aims to determine the shape and dimension of dental arches from a lingual perspective, and determine shape and size used for lingual Orthodontics.

DETAILED DESCRIPTION:
The study sample comprised 70 Caucasian Brazilian individuals with normal occlusion and at least four of Andrew's six keys. Maxillary and mandibular dental casts were digitized (3D) and the images were analyzed by Delcam Power SHAPET 2010 software. Landmarks on the lingual surface of teeth were selected to determine the shape and size of dental arches.

ELIGIBILITY:
Inclusion Criteria:criterion was that individuals should be at least 15 years of age all permanent teeth in occlusion -

Exclusion Criteria:with no odontogenic abnormalities

-

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 70 Caucasian Brazilian individuals (28 men and 42 women) with an average age of 16.4 years
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Statistic study | six months
  describe arch form similar a mushroom arch

CONTACTS AND LOCATIONS:
Overall Officials: Shirley SN Pignatari, PHD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Disciplina de Otorrinolaringologia Pediatrica, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
The 70 pairs of cast models were digitized with a 3D Dental Wings™ Scanner (model DW5-140, Montreal, Quebec, Canada). Images were analyzed by Delcam Power SHAPE™ software (2010, Birmingham, UK).

REFERENCES:
- [Result] Lombardo L, Saba L, Scuzzo G, Takemoto K, Oteo L, Palma JC, Siciliani G. A new concept of anatomic lingual arch form. Am J Orthod Dentofacial Orthop. 2010 Sep;138(3):260.e1-260.e13; discussion 260-1. doi: 10.1016/j.ajodo.2010.04.022. PMID 20816292